CLINICAL TRIAL: NCT00423800
Title: Efficacy and Safety of 24 vs 48 Weeks of Pegetron® (Peginterferon Alfa-2b + Ribavirin) Therapy (1.5 mcg/kg/Week + 800-1200 mg/Day) in Naïve Genotype 1 Hepatitis C Patients With High Baseline Viral Load Who Are HCV-RNA Negative at Week 4 and Week 12
Brief Title: Efficacy and Safety of 24 vs 48 Weeks of Pegetron® (Peginterferon Alfa-2b + Ribavirin) in Naïve Genotype 1 Hepatitis C (Study P05016)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to difficulty in recruiting participants.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05016
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2b; Powders; Solutions; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegetron® - 24 Weeks (Experimental): Participants are treated with Pegetron® (pegylated interferon alfa-2b and ribavirin) for 8 weeks and then randomized to an additional 16 weeks of treatment
  Interventions: Drug: Combination of pegylated interferon alfa-2b (PEG) and ribavirin (RBV)
- Pegetron®- 48 Weeks (Active Comparator): Participants are treated with Pegetron® (pegylated interferon alfa-2b and ribavirin) for 8 weeks and then randomized to an additional 40 weeks of treatment.
  Interventions: Drug: Combination of pegylated interferon alfa-2b (PEG) and ribavirin (RBV)

INTERVENTIONS:
Drug: Combination of pegylated interferon alfa-2b (PEG) and ribavirin (RBV) — 1. Powder for Solution in Redipen® (pegylated interferon alfa-2b) (80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 24 or 48 weeks
  2. 200 mg ribavirin capsules, oral, weight-based dose of 800, 1000, or 1200 mg, daily for up to 24 or 48 weeks
  Other Names: PEGETRON® combination therapy; (a) SCH 54031, PEGETRON® (peginterferon alfa-2b) Powder for Solution; (b) SCH 18908, PEGETRON® (ribavirin) Capsules

SUMMARY:
This is a Phase IIIB randomized, controlled, multi-centre, open-label study of 24 versus 48 weeks therapy with Pegetron® (peginterferon alfa-2b + ribavirin) at standard doses in naïve Hepatitis C Virus (HCV) genotype 1 high viral load (HVL) participants who are Hepatitis C Virus-Ribonucleic Acid (HCV-RNA) negative at Week 4. HVL will be defined as HCV-RNA of >600,000 IU/mL prior to the initiation of therapy. Participants with genotype 1 baseline HVL prescribed Pegetron® (peginterferon and ribavirin) in the usual manner in accordance with the marketing authorization and who are viral negative at Week 4 will be randomized at Week 8 to receive a total of 24 or 48 weeks of therapy. Participants will be required to have their baseline and Week-12 viral load analyzed by the same local laboratory using the standard of care test used by the site. Qualitative testing at Week 4, 8, 16-20, 24, and 48 may be conducted either by local laboratory or a central laboratory identified by the sponsor using an assay specified by the sponsor. No additional interventions outside of the clinic's standard of care and the conditions of the Canadian product monograph for Pegetron® will be applied to participants.

ELIGIBILITY:
Inclusion Criteria:

* Must demonstrate willingness to participate in the study.
* Diagnosed with chronic HCV.
* Between 18 and 65 years of age of either gender and of any race.
* a. HCV positive, >600,000 IU/mL at baseline AND b. Genotype 1.
* Suitable for treatment with Pegetron® per the Canadian product monograph.
* Investigator has already decided to treat with PEGETRON REDIPEN®

1.5mcg/kg/week of peginterferon alpha-2b plus 800-1200 mg /day of ribavirin.

* HCV-RNA negative at treatment week 4.
* Meet certain minimum laboratory values at the week 4 screening visit.
* Women of childbearing potential and male partners must agree to use a medically accepted method of contraception prior to screening, while receiving protocol-specified medication, and for 6 months after stopping the medication. Acceptable methods of contraception include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD, oral or injectable hormonal contraceptive, and surgical sterilization (e.g. hysterectomy or tubal ligation).

Exclusion Criteria:

* Had previous interferon-based therapy for Chronic Hepatitis C.
* Active Hepatitis B virus (HBV) infection.
* Human Immunodeficiency Virus (HIV) antibody positive.
* Cirrhotic (Stage 4 on Metavir system).
* Uncontrolled history or current severe depression or psychoses.
* Uncontrolled epilepsy.
* Use of illicit drugs.
* History of non-compliance to medical regimens.
* Liver disease other than from chronic hepatitis C.
* Participating in any other clinical study.
* Used any investigational drugs within 30 days of screening.
* Participants weighing < 40 kg or > 125 kg.
* Pregnant women or women who plan to become pregnant or sexual partners of women who want to become pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 participants were enrolled. 51 participants were screening failures, were not randomized and are not included in the study. Of the 5 participants randomized, 2 did not meet inclusion/exclusion criteria. All 5 are included in the intent-to-treat (ITT) population.
Groups:
- Pegetron® - 24 Weeks: Participants are treated for 8 weeks and then randomized to an additional 16 weeks of treatment
- Pegetron® - 48 Weeks: Participants are treated for 8 weeks and then randomized to an additional 40 weeks of treatment
Period: Overall Study
Arm/Group | Pegetron® - 24 Weeks | Pegetron® - 48 Weeks
Started | 3 | 2
Completed | 3 | 1
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegetron® - 24 Weeks | Pegetron® - 48 Weeks | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (9.5) | 22 (0) | 41.2 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Sustained Virologic Response
Description: Participants were tested for the presence of Hepatitis C Virus-Ribonucleic Acid (HCV-RNA) in blood by Qualitative Polymerase Chain Reaction (qPCR). If the HCV-RNA is not detectable, the participant is negative for HCV-RNA.
  Sustained virologic responders were participants negative for HCV-RNA at 24 weeks following the completion of therapy. A Participant that withdrew prior to 24 weeks following the completion of therapy was considered a non-responder.
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Measure: Number; unit: Participants
Arm/Group | Pegetron® - 24 Weeks | Pegetron® - 48 Weeks
Number analyzed (Participants) | 3 | 2
Participants
  Responders | 3 | 1
  Non-responders | 0 | 1

2. Secondary Outcome: Number of Participants With a Virological Relapse
Description: Participants were tested for the presence of Hepatitis C Virus-Ribonucleic Acid (HCV-RNA) in blood by Qualitative Polymerase Chain Reaction (qPCR).
  Virological relapse in participants was defined as having negative virology (HCV-RNA) at end of treatment, but positive virology (HCV-RNA) again at 24 weeks of follow up post treatment.
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: ITT population that completed the study.
Measure: Number; unit: Participants
Arm/Group | Pegetron® - 24 Weeks | Pegetron® - 48 Weeks
Number analyzed (Participants) | 3 | 1
Participants
  Participants with Virological Relapse | 0 | 0
  Participants with No Virological Relapse | 3 | 1

ADVERSE EVENTS:
Description: Included are the adverse events (AEs) for all randomized participants (Pegetron® - 24 weeks and Pegetron® - 48 weeks). Also included are two (2) Serious Adverse Events (SAEs) for 2 participants on commercial Pegetron® who were screen fails for this study and were never randomized (Screen Failures).
Groups:
- Screen Failures: Two participants on commercial Pegetron® who were screen fails and were never randomized had SAEs. Both SAEs were are reported here.
- Pegetron® - 24 Weeks: Participants are treated for 8 weeks with Pegetron® and then randomized to an additional 16 weeks of treatment.
- Pegetron® - 48 Weeks: Participants are treated for 8 weeks with Pegetron® and then randomized to an additional 40 weeks of treatment.
Arm/Group | Screen Failures | Pegetron® - 24 Weeks | Pegetron® - 48 Weeks
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 2/3 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screen Failures (N=2) | Pegetron® - 24 Weeks (N=3) | Pegetron® - 48 Weeks (N=2)
GROIN ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIC SEIZURE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screen Failures (N=2) | Pegetron® - 24 Weeks (N=3) | Pegetron® - 48 Weeks (N=2)
EYE IRRITATION (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
CHILLS (General disorders) | 0 (0) | 1 (2) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 2 (3) | 0 (0)
IRRITABILITY (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 2 (4) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
AFFECT LABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the small sample size (n=5), no conclusions should be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 45 days from the time submitted to the sponsor for review.